CLINICAL TRIAL: NCT04046406
Title: Pelvic Pain Treated With MR-guided Cryoanalgesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There were issues with equipment and team fell apart due to departure of some members from the institution.
Sponsor: Johns Hopkins University (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00222178
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Pelvic Pain Syndrome; Groin Pain; Meralgia Paresthetica; Low Back Pain; Perineal Neuralgia
MeSH Terms: conditions — Femoral Neuropathy; Low Back Pain; Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pelvic pain syndromes (Experimental): Patients with pelvic pain syndromes who will undergo MR neurography-guided cryoanalgesia
  Interventions: Device: MR neurography-guided cryoanalgesia

INTERVENTIONS:
Device: MR neurography-guided cryoanalgesia — Treatment will be performed using a FDA-approved Galil Medical cryoablation system and FDA-approved Galil Medical cryoablation needles.

SUMMARY:
Pelvic pain syndromes have a high prevalence of up to 8% in the general population and up to 50% following pelvic trauma and pelvic surgery. While medical management is the initial therapeutic step, it is often ineffective with surgical decompression and resection of the putative nerves being the ultima ratio. Cryoablation can induce long-lasting nerve conduction blocks with resultant pain relief for several months. The objective of this study is to evaluate the effectiveness of magnetic resonance (MR) neurography-guided cryoanalgesia for the treatment of pelvic and associated pain syndromes.

DETAILED DESCRIPTION:
Pelvic pain syndromes including meralgia paresthetica, inguinodynia, and deep gluteal syndrome and others, which are caused by nerves including the the lateral femoral cutaneous nerve (LFCN), genitofemoral nerve (GFN), ilioinguinal nerve (IIN), iliohypogastric nerve (IHN), pudendal nerve (PN), obturator nerve (ON), posterior femoral cutaneous nerve (PFCN), and others, have a high prevalence of up to 8% in the general population and up to 50% following pelvic trauma and pelvic surgery, including episiotomy, orthopedic instrumentation and surgical hernia repair. While medical management is the initial therapeutic step, it is often ineffective with surgical decompression and resection of the putative nerves being the ultima ratio. Cryoablation of sensory nerves at temperatures of approximately 40 degrees Celsius and below (Cryoanalgesia) can induce long-lasting nerve conduction blocks with resultant pain relief for several months, which could be an effective treatment option for a large number of patients in this group before, instead of, and after failed surgical treatment. Cryoablation affords several advantages over other thermal or chemical ablation techniques, including direct visualization of the ablation zone, decreased intraprocedural and postprocedural pain, and the ability to simultaneously use multiple probes in variable configurations to create tailored additive overlapping ablation zones. In contrast to surgical or heat-mediated ablation, cryoablation does not disrupt the acellular epineurium or perineurium, which reduces the risk of neuroma formation and may allow eventual nerve regeneration, after which the cryoanalgesia can be repeated. Interventional MR neurography at 3 Tesla describes the combined use of high-resolution MRI for the visualization of smallest nerves that are located deep inside the pelvis, targeting, placement of needles and probes, and process monitoring, such as growth of the ice ball and relationship to the target nerves. The use of interventional MR neurography is thus ideally suited to perform cryoanalgesia with the highest technical accuracy and safety. The objective of this study is to evaluate the effectiveness of MR neurography-guided cryoanalgesia for the treatment of pelvic and associated pain syndromes.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 100 years
* Chronic pelvic pain for at least 3 months and no adequate pain relief defined as persistent worst pain 4 or above on an 11-point visual analogue scale of 0 (no pain) to 10 (pain as bad as subject can imagine) despite conservative treatments, including but not limited to oral pain medication including NSAIDs and narcotics, physical therapy, and nerve block.
* The 'worst pain' must be reported to be 4 or above on an 11-point visual analogue scale of 0 (no pain) to 10 (pain as bad as subject can imagine)
* Pain must be from a single lumbosacral nerves confirmed with selective nerve blocks providing adequate temporary pain. The selectivity of the nerve block will be confirmed on MR images documenting that the injected local anesthetic immerses the targeted nerve and that there is absence of spread of local anesthetic to adjacent nerves to exclude confounding anesthesia. Adequate pain relief will be defined by pain relief of greater 50% after the nerve block and rest and with aggravating exercise.
* The target nerve is amenable to cryoablation with MRI guidance
* Cryoablation should be performed within 3 months of the nerve block
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up
* Known coagulopathy or bleeding disorders are controlled

Exclusion Criteria:

* Confounding pain syndromes or conditions.
* Previous nerve surgery
* Currently pregnant, nursing, or wishing to become pregnant during the study
* Serious medical illness, including any of the following: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction, cerebrovascular event within 6 months prior to the screening visit
* Concurrent participation in other studies that could affect the primary endpoint

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in self-reported average pain score | Baseline and 12 weeks post cryoablation procedure
  Therapeutic success is defined as 50 percent or more pain reduction and/or an absolute pain level below 2 on an 11-point visual analog pain scale of 0 (no pain) to 10 (pain as bad as subject can imagine).

SECONDARY OUTCOMES:
Change in pain intensity as assessed by the Brief Pain Inventory (BPI) | Baseline, 1, 3, 6, 9, 12, and 18 months post cryoablation procedure
  This test will assess pain intensity (worst pain, least pain, average pain, pain right now) measured on an 11-point visual analogue scale of 0 (no pain) to 10 (pain as bad as subject can imagine).
Change in percentage pain relief | Baseline, 1, 3, 6, 9, 12, and 18 months post cryoablation procedure
  This test will assess percentage pain relief since baseline on an 11-point visual analogue scale with 10 percent increments with higher scores indicating more relief.
Change in analgesic medication use | Baseline, 1, 3, 6, 9, 12, and 18 months post cryoablation procedure
  This test will assess analgesic medication use in order to assess change in analgesic medications by recording the daily dose and type of medication. Morphine Equivalent Daily Dosing and Comparable NSAID Dose Levels will be used to compare the dose of different pain medications.
Change in pain interference as assessed by the BPI | Baseline, 1, 3, 6, 9, 12, and 18 months post cryoablation procedure
  This test will assess pain interference using a 7-item questionnaire on the BPI (that includes general activity, mood, walking ability, normal walk, relations with other people, sleep, and enjoyment of life) scored on an 11-point visual analogue scale from 0 to 10 with 0 meaning no interference and 10 meaning complete interference.
Change in Self-Assessment of Treatment as assessed by a 5-item questionnaire | Baseline, 1, 3, 6, 9, 12, and 18 months post cryoablation procedure
  The change in the self-assessment of the treatment offered patients will be assessed with a 5-item questionnaire that is graded on a 5-point Likert scale which ranges from -2 to +2 with positive scores indicating better satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fritz, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No